CLINICAL TRIAL: NCT06919887
Title: Evaluation of a Mobile Phone Application Tool for Menopause Symptom Management
Brief Title: A Randomized Controlled Trial of Menopausal Tool/App for Women
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephanie Faubion, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-013662
Record Dates: First submitted 2025-03-25; First posted 2025-04-09 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Menopausal Symptoms; Menopause Symptom Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The tool/app, EMMII by BettrHealth (Experimental): EMMII by BettrHealth Technology consists of educational components designed to enable women to more effectively identify menopause symptoms and feel confident in seeking treatment to address their symptoms
  Interventions: Other: EMMII
- Comparison Group/ Control Group (Experimental): Patients will receive the Mayo Clinic Patient Education Pamphlet MC5544 "Perimenopause & Menopause".
  Interventions: Other: Comparison Group

INTERVENTIONS:
Other: EMMII — The tool/app, consists of educational components designed to enable women to more effectively identify menopause symptoms and feel confident in seeking treatment to address their symptoms. The tool/app also produces a tailored menopause discussion guide for patients to bring to their primary care appointment.
  Arms: The tool/app, EMMII by BettrHealth
Other: Comparison Group — Receive educational menopause pamphlet describing menopause symptoms and evidence-based treatment options.
  Arms: Comparison Group/ Control Group

SUMMARY:
The purpose of this study is about assessing the utilization of a mobile phone application (app), designed to improve the menopause experience of midlife women experiencing related symptoms and its association with menopause-related health care utilization

ELIGIBILITY:
For Patient Enrollment:

Inclusion Criteria:

* Women between the ages of 45 and 55
* English speaking (app only available in English)
* Able to provide informed consent
* Experiencing menopause symptoms, which will be assessed by a Menopause Rating Scale (MRS) survey score of ≥ 5
* Has an upcoming Mayo Clinic primary care appointment within 3 weeks of the enrollment and the MRS survey

Exclusion Criteria:

* Lack of willingness to engage with app
* Inability to provide informed consent

Ages: 24 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of app logins among intervention group. | Up to 6 weeks
Compare differences in rates of menopause treatment among intervention and comparison groups. | Up to 6 weeks
Mean score on a validated survey assessing perceived importance and availability of healthcare services for women's health conditions/concerns related to menopause | through study completion, an average of 1 year
Percentage of healthcare professionals reporting 'high' & 'low' confidence in diagnosing and managing menopause symptoms | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
To uphold the informed consent agreements with participants, which may have specified restrictions on data sharing beyond the study team

REFERENCES:
- [Derived] Karam J, Paul MM, Shufelt C, Ravikumar P, Fratianni AM, Oloyede S, Pagel EM, Hedges MS, Kapoor E, Kling JM, Cole K, Chaudhry R, Faubion SS. Evaluating the Efficacy of a Mobile Phone App in Enhancing Menopause Knowledge and Shared Decision-Making: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Oct 8;14:e76536. doi: 10.2196/76536. PMID 41061260